CLINICAL TRIAL: NCT05026307
Title: Corneal Topographic Changes After Pterygium Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Abdelraheem, Principle investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-06-03
Record Dates: First submitted 2021-08-22; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pterygium (Experimental): Simple surgical excision of pterygium withe bare sclera
  Interventions: Procedure: Excision of pterygium

INTERVENTIONS:
Procedure: Excision of pterygium — Simple surgical excision of pterygium with bare sclera

SUMMARY:
The purpose of the study is to assess the corneal topographic changes after primary pterygium surgery

DETAILED DESCRIPTION:
Prospective interventional comparative study . This study will be conducted on eyes with primary pterygium before and after successful excision in department of ophthalmology, Sohag university hospital to assess the corneal topographic changes using pentacam .

Postoperative evaluation will be scheduled for one month ,three and six months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary pterygium

Exclusion Criteria:

* patients with recurrent pterygium
* patients with primary pterygium with other ocular pathologies.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Changes in corneal topography | One month, three and six months postoperative
  Detection of changes in corneal topography using Pentacam

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nangia V, Jonas JB, Nair D, Saini N, Nangia P, Panda-Jonas S. Prevalence and associated factors for pterygium in rural agrarian central India. The central India eye and medical study. PLoS One. 2013 Dec 4;8(12):e82439. doi: 10.1371/journal.pone.0082439. eCollection 2013. PMID 24324789
- [Background] Moran DJ, Hollows FC. Pterygium and ultraviolet radiation: a positive correlation. Br J Ophthalmol. 1984 May;68(5):343-6. doi: 10.1136/bjo.68.5.343. PMID 6712914
- [Background] Di Girolamo N, Chui J, Coroneo MT, Wakefield D. Pathogenesis of pterygia: role of cytokines, growth factors, and matrix metalloproteinases. Prog Retin Eye Res. 2004 Mar;23(2):195-228. doi: 10.1016/j.preteyeres.2004.02.002. PMID 15094131
- [Background] Xu Z, Li W, Jiang J, Zhuang X, Chen W, Peng M, Wang J, Lu F, Shen M, Wang Y. Characteristic of entire corneal topography and tomography for the detection of sub-clinical keratoconus with Zernike polynomials using Pentacam. Sci Rep. 2017 Nov 28;7(1):16486. doi: 10.1038/s41598-017-16568-y. PMID 29184086